CLINICAL TRIAL: NCT02268461
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) Treatment of Post-Stroke Spasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1408M53261
Record Dates: First submitted 2014-09-09; First posted 2014-10-20 (Estimated); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Spasticity
Keywords: Post-Stroke Spasticity
MeSH Terms: conditions — Muscle Spasticity | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- rTMS then Sham rTMS (Active Comparator): repetitive Transcranial Magnetic Stimulation (rTMS)
  Interventions: Device: repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham rTMS then Real rTMS (Sham Comparator): Sham repetitive Transcranial Magnetic Stimulation (Sham rTMS)
  Interventions: Device: Sham repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation (rTMS) — The treatment arm will consist of 3 daily treatment sessions. One treatment session in this study with real rTMS will consist of 600 pulses of 1Hertz rTMS at an intensity of 90% of resting motor threshold (duration 10 minutes) applied to the primary motor area of the contralesional hemisphere.
  Other Names: Magstim 200^2 Magnetic Stimulator (MODEL 3010-00); Magstim Rapid^2 Magnetic Stimulator (MODE 3004-000)
  Arms: rTMS then Sham rTMS
Device: Sham repetitive Transcranial Magnetic Stimulation — Sham rTMS utilizes a coil that produces identical noise and tactile sensation to the real coil, but does not emit a magnetic field (0% intensity). Duration and frequency of auditory and tactile stimulation will be identical to the real intervention.
  Arms: Sham rTMS then Real rTMS

SUMMARY:
Spasticity is a common complication of stroke affecting quality of life. Spasticity involves exaggerated stretch reflexes that create stiffness in muscles with associated loss of motion and functional control. Traditional treatments involve range of motion, medications, and sometimes surgery. Each of these has its own limitations, which has invited exploration of alternative modes of treatment. One such treatment with the potential to benefit spasticity is repetitive Transcranial Magnetic Stimulation (rTMS).

The purpose of this study is to determine whether patients with upper limb spasticity as a consequence of a chronic stroke can benefit from stimulation of the non-affected hemisphere of the brain with low-frequency (inhibitory) repetitive Transcranial Magnetic Stimulation (rTMS), potentially leading to a reduction of spasticity and clinical improvement in upper limb function.

DETAILED DESCRIPTION:
The purpose of this pilot study is to evaluate the efficacy of rTMS versus placebo for spasticity reduction in a cross-over design in 6 people with stroke.

Our research question is: In patients with upper extremity spasticity as a consequence of chronic stroke, does stimulation of the contralesional motor cortex with low-frequency (inhibitory) rTMS lead to reduction of spasticity and thereby clinical improvement in upper extremity function? Our rationale is that the pathophysiology of post-stroke spasticity is primarily driven by ensuant cortical derangement, and further, that this derangement can be mitigated to a clinically meaningful extent by proper utilization of rTMS directed at these foci. Optimized rTMS treatment protocols may even achieve efficacy that surpasses current mainstays of spasticity management.

Patients will be randomly assigned to receive either rTMS or placebo during their first treatment arm and then cross-over to receive the opposite treatment at the second treatment arm. A washout period of one month will occur between treatment arms. Each treatment arm will consist of 3 daily treatment sessions. Participants will present on a Monday for the pre-test assessment, Tuesday-Thursday for the treatment sessions and Friday for the post-test assessment. One treatment session will consist of 600 pulses of 1Hertz rTMS at an intensity of 90% of resting motor threshold (duration 10 minutes) applied to the primary motor area of the contralesional hemisphere. Sham rTMS intensity will be 0% but with a similar sound and scalp sensation. Assessments will be made at each session, and will be conducted at pre-test, post-test, and one-month follow-up. The one month follow-up test will serve as the pretest for the next treatment arm. That is, after follow-up, patients will cross-over to receive the opposite treatment in the same format. Safety has already been demonstrated for our protocol. Data will be analyzed with methods appropriate to a single-subject crossover design (visual analysis, confidence intervals and 2-Standard Deviation bandwidth).

The primary outcome that we will measure is reduction of spasticity at the fingers and wrist. A secondary outcome of interest is functional improvement of the spastic upper limb.

ELIGIBILITY:
Inclusion Criteria:

1. first-time stroke
2. stroke at least six months prior to onset of study with chronic sequela of spasticity
3. stroke location- either cortical or subcortical
4. stroke type- either hemorrhagic or ischemic
5. stroke hemisphere- either left or right, dominant or non- dominant hemisphere
6. 18 years of age or older
7. gender- either male or female
8. ability to follow three-step directions
9. demonstration of 10 degrees of active extension at the metacarpophalangeal joint and wrist of the paretic upper extremity
10. demonstration of consistent resting motor evoked potential from ipsilesional and contralesional hemispheres
11. sufficient ambulation or wheelchair mobility to allow subject to present to treatment and testing areas with minimum assist

Exclusion Criteria:

1. history of seizure within the past two years
2. inability to follow three-step directions
3. anosognosia
4. moderate to severe receptive aphasia
5. inability to give informed consent
6. premorbid spasticity or neurologic impairment prior to stroke
7. co-morbidities impairing upper extremity function such as fracture or deformity
8. indwelling metal or medical devices incompatible with TMS
9. pregnancy
10. bi-hemispheric or multifocal stroke
11. dementia
12. neurolytic injection within the 3 months prior to onset of study or planned neurolytic injection during study period
13. planned vacation or travel during study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-12; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Timp, DO, Principal Investigator — University of Minnesota, Physical Medicine and Rehabilitation; James R Carey, PhD, PT, Study Chair — University of Minnesota, Program in Physical Therapy; Florence S John, MD, MPH, Study Director — University of Minnesota, Physical Medicine and Rehabilitation; Kate Frost, MS, Study Director — University of Minnesota, Program in Physical Therapy
Locations (1):
- University of Minnesota, Clinical and Translational Science Institute, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Carmichael ST, Tatsukawa K, Katsman D, Tsuyuguchi N, Kornblum HI. Evolution of diaschisis in a focal stroke model. Stroke. 2004 Mar;35(3):758-63. doi: 10.1161/01.STR.0000117235.11156.55. Epub 2004 Feb 12. PMID 14963280
- [Background] Duque J, Murase N, Celnik P, Hummel F, Harris-Love M, Mazzocchio R, Olivier E, Cohen LG. Intermanual Differences in movement-related interhemispheric inhibition. J Cogn Neurosci. 2007 Feb;19(2):204-13. doi: 10.1162/jocn.2007.19.2.204. PMID 17280510
- [Background] Murase N, Duque J, Mazzocchio R, Cohen LG. Influence of interhemispheric interactions on motor function in chronic stroke. Ann Neurol. 2004 Mar;55(3):400-9. doi: 10.1002/ana.10848. PMID 14991818
- [Background] Kirton A, Chen R, Friefeld S, Gunraj C, Pontigon AM, Deveber G. Contralesional repetitive transcranial magnetic stimulation for chronic hemiparesis in subcortical paediatric stroke: a randomised trial. Lancet Neurol. 2008 Jun;7(6):507-13. doi: 10.1016/S1474-4422(08)70096-6. Epub 2008 May 1. PMID 18455961
- [Background] Grefkes C, Nowak DA, Wang LE, Dafotakis M, Eickhoff SB, Fink GR. Modulating cortical connectivity in stroke patients by rTMS assessed with fMRI and dynamic causal modeling. Neuroimage. 2010 Mar;50(1):233-42. doi: 10.1016/j.neuroimage.2009.12.029. Epub 2009 Dec 18. PMID 20005962
- [Background] Burn J, Dennis M, Bamford J, Sandercock P, Wade D, Warlow C. Epileptic seizures after a first stroke: the Oxfordshire Community Stroke Project. BMJ. 1997 Dec 13;315(7122):1582-7. doi: 10.1136/bmj.315.7122.1582. PMID 9437276
- [Background] Carey JR, Kimberley TJ, Lewis SM, Auerbach EJ, Dorsey L, Rundquist P, Ugurbil K. Analysis of fMRI and finger tracking training in subjects with chronic stroke. Brain. 2002 Apr;125(Pt 4):773-88. doi: 10.1093/brain/awf091. PMID 11912111
- [Background] Carey JR, Evans CD, Anderson DC, Bhatt E, Nagpal A, Kimberley TJ, Pascual-Leone A. Safety of 6-Hz primed low-frequency rTMS in stroke. Neurorehabil Neural Repair. 2008 Mar-Apr;22(2):185-92. doi: 10.1177/1545968307305458. Epub 2007 Sep 17. PMID 17876070
- [Background] Kakuda W, Abo M, Momosaki R, Yokoi A, Fukuda A, Ito H, Tominaga A, Umemori T, Kameda Y. Combined therapeutic application of botulinum toxin type A, low-frequency rTMS, and intensive occupational therapy for post-stroke spastic upper limb hemiparesis. Eur J Phys Rehabil Med. 2012 Mar;48(1):47-55. Epub 2011 Nov 9. PMID 22071503
- [Background] Kakuda W, Abo M, Kobayashi K, Momosaki R, Yokoi A, Fukuda A, Ito H, Tominaga A, Umemori T, Kameda Y. Anti-spastic effect of low-frequency rTMS applied with occupational therapy in post-stroke patients with upper limb hemiparesis. Brain Inj. 2011;25(5):496-502. doi: 10.3109/02699052.2011.559610. PMID 21456998
- [Background] Kakuda W, Abo M, Kobayashi K, Momosaki R, Yokoi A, Fukuda A, Ishikawa A, Ito H, Tominaga A. Low-frequency repetitive transcranial magnetic stimulation and intensive occupational therapy for poststroke patients with upper limb hemiparesis: preliminary study of a 15-day protocol. Int J Rehabil Res. 2010 Dec;33(4):339-45. doi: 10.1097/MRR.0b013e32833cdf10. PMID 20613547
- [Background] Kirton A, Deveber G, Gunraj C, Chen R. Cortical excitability and interhemispheric inhibition after subcortical pediatric stroke: plastic organization and effects of rTMS. Clin Neurophysiol. 2010 Nov;121(11):1922-9. doi: 10.1016/j.clinph.2010.04.021. PMID 20537584
- [Background] Kujirai T, Caramia MD, Rothwell JC, Day BL, Thompson PD, Ferbert A, Wroe S, Asselman P, Marsden CD. Corticocortical inhibition in human motor cortex. J Physiol. 1993 Nov;471:501-19. doi: 10.1113/jphysiol.1993.sp019912. PMID 8120818
- [Background] Liepert J, Storch P, Fritsch A, Weiller C. Motor cortex disinhibition in acute stroke. Clin Neurophysiol. 2000 Apr;111(4):671-6. doi: 10.1016/s1388-2457(99)00312-0. PMID 10727918
- [Background] Mally J, Dinya E. Recovery of motor disability and spasticity in post-stroke after repetitive transcranial magnetic stimulation (rTMS). Brain Res Bull. 2008 Jul 1;76(4):388-95. doi: 10.1016/j.brainresbull.2007.11.019. Epub 2007 Dec 26. PMID 18502315
- [Background] Mathiowetz V, Volland G, Kashman N, Weber K. Adult norms for the Box and Block Test of manual dexterity. Am J Occup Ther. 1985 Jun;39(6):386-91. doi: 10.5014/ajot.39.6.386. PMID 3160243
- [Background] Mathiowetz V, Federman S, Wiemer, D. Box and Block Test of Manual Dexterity: Norms for 6-19 Year Olds. CJOT. 1985b; 52(5): 241-245.
- [Background] McDonnell MN, Orekhov Y, Ziemann U. The role of GABA(B) receptors in intracortical inhibition in the human motor cortex. Exp Brain Res. 2006 Aug;173(1):86-93. doi: 10.1007/s00221-006-0365-2. Epub 2006 Feb 18. PMID 16489434
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Soliman EZ, Sorlie PD, Sotoodehnia N, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2012 update: a report from the American Heart Association. Circulation. 2012 Jan 3;125(1):e2-e220. doi: 10.1161/CIR.0b013e31823ac046. Epub 2011 Dec 15. No abstract available. PMID 22179539
- [Background] Sommerfeld DK, Gripenstedt U, Welmer AK. Spasticity after stroke: an overview of prevalence, test instruments, and treatments. Am J Phys Med Rehabil. 2012 Sep;91(9):814-20. doi: 10.1097/PHM.0b013e31825f13a3. PMID 22760104
- [Background] Theilig S, Podubecka J, Bosl K, Wiederer R, Nowak DA. Functional neuromuscular stimulation to improve severe hand dysfunction after stroke: does inhibitory rTMS enhance therapeutic efficiency? Exp Neurol. 2011 Jul;230(1):149-55. doi: 10.1016/j.expneurol.2011.04.010. Epub 2011 Apr 16. PMID 21524650
- [Background] Wassermann EM, Wedegaertner FR, Ziemann U, George MS, Chen R. Crossed reduction of human motor cortex excitability by 1-Hz transcranial magnetic stimulation. Neurosci Lett. 1998 Jul 10;250(3):141-4. doi: 10.1016/s0304-3940(98)00437-6. PMID 9708852
- [Background] Weiduschat N, Thiel A, Rubi-Fessen I, Hartmann A, Kessler J, Merl P, Kracht L, Rommel T, Heiss WD. Effects of repetitive transcranial magnetic stimulation in aphasic stroke: a randomized controlled pilot study. Stroke. 2011 Feb;42(2):409-15. doi: 10.1161/STROKEAHA.110.597864. Epub 2010 Dec 16. PMID 21164121
- [Background] Braddom, Randall L., Ralph M. Buschbacher. Ch 30 Spasticity Management. Physical Medicine & Rehabilitation. Saunders Elsevier 2007; 641-55.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | rTMS Then Sham rTMS | Sham rTMS Then Real rTMS
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rTMS Then Sham rTMS | Sham rTMS Then Real rTMS | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Data was not collected Population: Data not collected
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Contralesional Corticospinal Excitability
Description: Motor evoked potentials (MEPs) were measured using surface EMG. The average amplitude of 10 MEPs measured at baseline was compared to the average of 10 MEPs measured at post-test and this difference is recorded as the change in corticospinal excitability. A greater negative value would indicate larger post-test MEPs and increased corticospinal excitability.
Time Frame: From Day 1 to Day 5
Measure: Mean (Standard Deviation); unit: microVolts
Groups:
- rTMS: repetitive Transcranial Magnetic Stimulation (rTMS)
  repetitive Transcranial Magnetic Stimulation (rTMS): The treatment arm will consist of 3 daily treatment sessions. One treatment session in this study with real rTMS will consist of 600 pulses of 1Hertz rTMS at an intensity of 90% of resting motor threshold (duration 10 minutes) applied to the primary motor area of the contralesional hemisphere.
- Real rTMS: Sham repetitive Transcranial Magnetic Stimulation (Sham rTMS)
  Sham repetitive Transcranial Magnetic Stimulation: Sham rTMS utilizes a coil that produces identical noise and tactile sensation to the real coil, but does not emit a magnetic field (0% intensity). Duration and frequency of auditory and tactile stimulation will be identical to the real intervention.
Arm/Group | rTMS | Real rTMS
Number analyzed (Participants) | 4 | 4
microVolts | 67.88 (384.91) | -37.23 (542.11)

2. Primary Outcome: Change From Baseline Finger Tracking Score
Description: An electrogoniometer attached to the hand was used to measure index finger movement. Patients tracked a sine wave that ranged from 85% to 15% of their individual max range of motion which does impact the accuracy measure scale. Accuracy of tracking along with the target waveform was assessed on a scale ranging from -100 to 100 (100 being perfect accuracy).
Time Frame: From Day 1 to Day 5
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Sham: Sham repetitive Transcranial Magnetic Stimulation (Sham rTMS)
  Sham repetitive Transcranial Magnetic Stimulation: Sham rTMS utilizes a coil that produces identical noise and tactile sensation to the real coil, but does not emit a magnetic field (0% intensity). Duration and frequency of auditory and tactile stimulation will be identical to the real intervention.
Arm/Group | rTMS | Sham
Number analyzed (Participants) | 4 | 4
score on a scale | 11.95 (29.65) | 8.01 (27.18)

3. Secondary Outcome: Change in Stroke Impact Scale
Description: Change from baseline stroke impact scale score The Stroke Impact Scale (SIS) is a standardized self-reported questionnaire used to assess the impact of stoke on an individual's quality of life.
  Scores range from 0-100 with higher scores indicating greater functionality and quality of life.
Time Frame: From Day 1 to Day 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rTMS | Sham
Number analyzed (Participants) | 4 | 4
score on a scale | -0.25 (0.433) | -0.5 (0.87)

4. Secondary Outcome: Change From Baseline Resting Motor Threshold
Description: Average change from baseline resting motor threshold The resting motor threshold (RMT) is the lowest possible stimulator output (% maximal stimulator output) required to reliably elicit a motor evoked potential. A lower RMT would indicate increased corticospinal excitability.
Time Frame: From Day 1 to Day 5
Measure: Mean (Standard Deviation); unit: %MSO
Arm/Group | rTMS | Sham
Number analyzed (Participants) | 4 | 4
%MSO | -2.25 (4.49) | -3.75 (12.6)

ADVERSE EVENTS:
Arm/Group | rTMS | Sham
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes